CLINICAL TRIAL: NCT02221180
Title: A Single-Dose, Open-Label, Randomized, 4-Way Crossover Pivotal Study to Assess the Bioequivalence of the Metformin Component of the Fixed Dose Combination Tablet of Canagliflozin and Metformin Immediate Release (IR) 1 x (150 mg/500 mg) With Respect to the Metformin IR Tablet (Locally Sourced From Canada [Glucophage, 1 x 500 mg]) Coadministered With Canagliflozin (1 x 50 mg and 1 x 100 mg) in Healthy Fed and Fasted Subjects
Brief Title: Bioequivalence Study of Metformin Component of Fixed Dose Combination (FDC) Immediate Release (IR) Tablet of Canagliflozin and Metformin Compared to Metformin IR Tablet Co-administered With Canagliflozin in Healthy Fed and Fasted Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR104980; 28431754DIA1071 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Bioequivalence
Keywords: Bioequivalence; Metformin; Canagliflozin; Healthy
MeSH Terms: interventions — Canagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence ABDC (Experimental): Treatment A (1 immediate release (IR) fixed dose combination [FDC] tablet containing canagliflozin 150 milligram [mg] and metformin 500 mg orally under fed condition) on Day 1 of treatment period 1, followed by Treatment B (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fed condition) on Day 1 of treatment period 2, followed by Treatment D (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fasted condition) on Day 1 of treatment period 3, then Treatment C (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fasted condition) on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Immediate Release (IR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin
- Treatment Sequence BCAD (Experimental): Treatment B (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fed condition) on Day 1 of treatment period 1, followed by Treatment C (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fasted condition) on Day 1 of treatment period 2, followed by Treatment A (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fed condition) on Day 1 of treatment period 3, then Treatment D (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fasted condition) on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Immediate Release (IR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin
- Treatment Sequence CDBA (Experimental): Treatment C (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fasted condition) on Day 1 of treatment period 1, followed by Treatment D (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fasted condition) on Day 1 of treatment period 2, followed by Treatment B (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fed condition) on Day 1 of treatment period 3, then Treatment A (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fed condition) on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Immediate Release (IR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin
- Treatment Sequence DACB (Experimental): Treatment D (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fasted condition) on Day 1 of treatment period 1, followed by Treatment A (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fed condition) on Day 1 of treatment period 2, followed by Treatment C (1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fasted condition) on Day 1 of treatment period 3, then Treatment B (1 canagliflozin tablet 50 mg and 1 canagliflozin tablet 100 mg along with 1 IR tablet of metformin 500 mg orally under fed condition) on Day 1 of treatment period 4. A washout period of 7 days will be maintained between each treatment period.
  Interventions: Drug: Canagliflozin and Metformin Immediate Release (IR) Fixed Dose Combination [FDC]; Drug: Canagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: Canagliflozin and Metformin Immediate Release (IR) Fixed Dose Combination [FDC] — Participants will receive 1 IR FDC tablet containing canagliflozin 150 mg and metformin 500 mg orally under fed or fasted condition in each treatment period as per treatment sequence.
  Other Names: CANA/MET IR FDC
Drug: Canagliflozin — Participants will receive canagliflozin 150 mg (50 mg+100 mg oral tablet) under fed or fasted condition in each treatment period as per treatment sequence.
  Other Names: CANA
Drug: Metformin — Participants will receive metformin 500 mg tablet orally under fed or fasted condition in each treatment period as per treatment sequence.
  Other Names: MET

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of metformin component of the canagliflozin and metformin immediate release (IR) fixed dose combination (FDC) tablet compared with the metformin IR tablet co-administered with canagliflozin in healthy fed and fasted participants.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label (identity of study drug will be known to volunteer and study staff), single-center, single-dose, 4-treatment, 4-way crossover (method used to switch participants from one study group to another in a clinical trial, like the flip of a coin) study in healthy adult participants. The study will have 3 phases: Screening Phase (approximately 3 weeks, Day -22 to Day -2), Open-Label Treatment Phase (consisting of 4 single-dose treatment periods of 3 days each [Day -1 to Day 2], each separated by a washout period of 7 days) and Follow-up Phase (5 to 7 days after last study-related procedure on Day 2 of treatment period 4). All the eligible participants will be randomly assigned to 1 of 4 treatment sequences and will receive 2 treatments under fasting and 2 treatments under fed conditions. Blood samples will be collected for evaluation of pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) at pre-dose and post-dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30 kilogram per square meter (kg/m^2) (inclusive) and a body weight of not less than 50 kg

Exclusion Criteria:

* History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Metformin | Pre-dose, up to 24 hours afterdose
  Plasma concentrations of metformin are used to evaluate how much metformin is in the blood over time.
Plasma Concentration of Canagliflozin | 2 hours after dosing
  Plasma concentrations of canagliflozin are used to evaluate how much canagliflozin is in the blood, 2 hours after dosing.

SECONDARY OUTCOMES:
Adverse Events | Up to approximately 58 days
  The number and type of adverse events will be reported from Day 1 of treatment period 1 through 5-7 days after treatment period 4 including a 7+/- 1 day washout period between treatment periods (total time is approximately 58 days).
Clinical Laboratory Test | Up to approximately 58 days
  Clinically relevant changes occurring in laboratory safety parameters will be evaluated.
Vital Signs | Up to approximately 58 days
  Blood pressure, pulse, and oral body temperature will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Lincoln, Nebraska, United States